CLINICAL TRIAL: NCT02153515
Title: Fingerprick Fresh Blood for Treatment of Chronic Corneal Ulcers, Persistent Epithelial Defects and Dry Eyes
Brief Title: Treating Dry Eyes and Corneal Ulcers With Fingerprick Autologous Blood
Acronym: FAB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bedford Hospital NHS Trust (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other); The Mater Infirmary Hospital Belfast, UK. (Unknown); Milton Keynes University Hospital NHS Foundation Trust (Other Government); Heart of England NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Birmingham Midland Eye Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 426/2014/340
Record Dates: First submitted 2014-05-02; First posted 2014-06-03 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Dry Eyes; Sjogren's Disease With Dry Eyes; Persistent Corneal Epithelial Defects; Chronic Corneal Ulcers
Keywords: Finger prick with diabetic lancet; Fingerprick; Fresh; Your own blood; autologous blood; Dry eyes; Sjogren's disease with dry eyes; Persistent corneal epithelial defects; Chronic corneal ulcers
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fingerprick of autologous blood (FAB) (Experimental): Fingerprick of autologous blood (FAB) four times a day for 2 months
  Interventions: Other: Your own ( autologous) finger prick of blood produced with a diabetic lancet

INTERVENTIONS:
Other: Your own ( autologous) finger prick of blood produced with a diabetic lancet

SUMMARY:
To investigate if fresh finger prick autologous blood (FAB) instead of serum from venesection, is a safe and effective treatment for dry eyes and corneal ulcers/ epithelial defects. Currently there are no studies on the use of whole fresh blood for the treatment of chronic ulcers, persistent epithelial defects or dry eyes. Unpublished case reports indicate that fresh blood can be an effective tool to the treatment of corneal pathology.

DETAILED DESCRIPTION:
Background Autologous serum is used for chronic ulcers and dry eyes. Currently there are no studies on the use of whole fresh blood for the treatment of chronic ulcers, persistent epithelial defects or dry eyes.

Dry eye syndrome (DES) refers to a common but highly heterogeneous group of ocular surface disorders with varying disease severity, due to lack of sufficient tears or sufficient quality of tears. Corneal and conjunctival studies, using a variety of definitions, have estimated the prevalence of ''significant'' DES to be about 10-20% in the adult population, although fortunately severe DES is less frequent (Hikichi et al., 1995; Bjerrum, 1997; Doughty et al., 1997; Bandeen-Roche et al., 1997; Caffery et al., 1998; McCarty et al., 1998; Schein et al., 1999; Moss et al., 2000; Begley et al., 2002; Chia et al., 2003; Lin et al., 2003; Schaumberg et al., 2003).

Dry eye is usually managed with conventional treatment of artificial tears, punctual plugs, occlusive goggles and bandage contact lenses. In spite of maximal conventional therapy, there is a cohort of patients who have persistent symptoms and signs. This represents a more serious ocular surface disorder with patients having significant visual impairment and disability. Particularly severe dry eye might be managed with contact lenses, botulinum toxin induced ptosis and surgical tarsorrhapy. These treatments are not without their own hazards such as infection from contact lenses, reduced vision from the ptosis or surgical tarsorrhapy, particularly in only seeing eyes.

Corneal ulcers are usually managed with artificial tears, antibiotic ointment, bandage contact lenses and steroids.

Autologous serum eye drops have been found in uncontrolled trials to be beneficial in these patients, improving the ocular surface and reducing symptoms (Poon et al., 2001; Fox et al., 1984; Tsubota et all, 1999;). In addition, impression cytology and in vitro toxicity testing demonstrated that serum drops have reduced toxicity compared with unpreserved hydroxypropylmethylcellulose (Noble et al., 2004; Poon et al., 2001)

Obtaining serum requires frequent venesection with significant amount of blood taken. It is also expensive. The serum is aliquoted into hundreds of bottles with the additional risk of bacterial contamination. It also requires a fridge and storage facilities for these aliquoted bottles at the patient's home. Because of these requirements some patients are excluded, for example patients with anaemia because they are unable to give blood. In addition, often there is a delay in starting the treatment for organizational and / or funding reasons that can be detrimental to the course of the disease, causing unnecessary surgery and corneal melt resulting in perforation with potential loss of the eye. The FAB method could be used immediately for patients who are awaiting conventional treatment for autologous blood. Furthermore it also appears that 100% autologous serum is more beneficial than 50% serum (Poon et al), thereby larger volumes of blood and/or more frequent venesection is required.

Autologous fresh blood is already used subconjunctivally to help heal leaking trabeculectomy blebs (Dinah et al.2010; Biswas et al. 2009; Burnstein et al. 2001; Haynes et al., 1999). Autologous blood is also used to help attach limbal autografts in cases of pterygium (de Wit et al. 2010) and in vitreoretinal macular hole surgery (Lai et al. 2009; Chuang et al. 2010; McCannel et al. 2008; Lai et al.,2005). No adverse effects have been reported in these studies. The object of this study is to investigate if serum via a drop of fresh blood is an effective treatment for dry eye and corneal ulcers which currently require venesected autologous blood and would be particularly useful in the current group of patients in whom venesection is contraindicated.

If shown to be effective this may replace current autologous serum practice and its ease of use and reduced cost may mean that it could be extended to other ocular surface diseases or moderate dry eyes and used earlier in corneal epithelial defects.

ELIGIBILITY:
Inclusion Criteria:

For Dry Eyes

* Patients with symptoms of dry eyes on at least QDS lubricants and who in addition:

  1. Satisfy at least one of the following criteria:

     Break up time (BUT) <5 seconds and Schirmer's test without anaesthesia <5 mm at 5 minutes OR presence of rose bengal /lissamine green or fluorescein staining of the ocular surface OR more than 80% score on OCI due to dry eyes (total score greater than or equal to 29/36)
  2. All patients must have unsuccessfully tried cyclosporine ointment or eye drops and temporary or permanent plugs or been offered punctual plugs and refused.

     For Corneal Ulceration
* Patients with epithelial defects of at least 2 weeks duration where conventional therapy failed. (Conventional therapy includes [if indicated] lubricants, antibiotic ointment, steroids and therapeutic contact lens wear)
* Any patient with an epithelial defect of at least 4 weeks' duration that has not completely healed with conventional therapy or who are refusing further conventional therapy. These patients would receive FAB therapy instead of tarsorrhaphy or botulinum toxin induced ptosis.

Exclusion Criteria:

* Fear of needles and unwillingness to carry out repeat finger pricks
* Infected finger or systemic infection or on systemic antibiotics for infection.
* Bleeding disorders and on warfarin anticoagulant therapy
* Epithelial defect was classified as a progressive corneal melt caused by an immunological process such as rheumatoid melt or Mooren's ulceration.
* Patients with active microbial infection, acute herpes simplex or herpes zoster keratitis, drug toxicity, vitamin A deficiency, or recurrent corneal erosion.
* Past Ophthalmic history of corneal transplantation.
* Pregnant or breast feeding women
* Children (under 16 years old).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Corneal ulcers / epithelial defects: Ulcers to heal within 4 weeks. Dry eyes: To improve signs (corneal and conjunctival staining, Schirmer's test, tear break up time ) or symptoms ( ocular comfort index questionnaire) | One month for corneal ulcers. Dry eyes 2 months.
  Follow ups are 3 days, 2 weeks , 4 weeks and 2 months after commencing treatment. Then again 1 month after stopping treatment.
  Criteria to stop treatment based on patient safety such as finger infection in protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Anant Sharma, FRCOphth, Study Chair — Moorfields Eye Hospital NHS Trust and Bedford Hospital NHS Trust
Locations (1):
- Moorfields Eye Centre at Bedford Hospital NHS Trust, Bedford, Bedfordshire, United Kingdom